CLINICAL TRIAL: NCT04929444
Title: Effectiveness of a Training Intervention to Improve the Approach of Patients With Vertigo in Primary Care. VERTAP Clinical Trial.
Brief Title: Training to Improve Vertigo Management in Primary Care
Acronym: VERTAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4R21/003; PI19/00736 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Vertigo; Vertigo, Paroxysmal
Keywords: primary care; vertigo; randomized clinical trial
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Intervention Model Description: Randomized community trial, by clusters (CG /IG), multicenter and open, taking as unit of allocation the primary care team (PCT). The professionals of the PCT that are in IG would receive the training at the beginning of the study and those of the control group will be offered after the conclusion of the same
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Active Comparator): The professionals of the primary care teams that are in Intervention group would receive the training at the beginning of the study
  Interventions: Other: Training on vertigo
- Common Practice (No Intervention): The professionals of the primary care teams that are in Control group will be offered the training after the conclusion of the study

INTERVENTIONS:
Other: Training on vertigo — Online training on vertigo management in primary care with a face-to-face session.
  On the one hand, the course will contain theoretical content and clinical cases will be used as the methodology of the course, with feedback paths for each correct or incorrect answer from the students and videos recorded expressly for the course. In addition, there will be a face-to-face session where all participants must perform the diagnostic and therapeutic maneuvers proposed in the course, to evaluate the use of the training and also to standardize the way of doing them for the study
  Arms: Training group

SUMMARY:
Objectives: To verify the effectiveness of a blended course in PC to improve adherence to clinical practice guidelines.

Design: randomized community trial, by clusters (control group -CG- / intervention group -IG-) Scope: 20 PCT (primary care teams)(10 per group) Outcome variables will be: Diagnostic records (proportion of nonspecific diagnoses such as dizziness and vertigo, with respect to specific diagnoses such as BPPV, vestibular neuritis); Derivations to otorhinolaryngologist (ENT) and neurologist; Prescription of antivertiginous medications and Number of days off work caused by vertigo-related.

Statistical analysis:Descriptive statistics of all the baseline variables will be carried out and, the differences between groups in the post-intervention outcome variables will be evaluated through the t-test. In the IG, a multivariate logistic regression model will identify response patterns based on the baseline variables of professionals and centers

DETAILED DESCRIPTION:
Vertigo is a prevalent pathology whose most frequent cause is benign paroxysmal positional vertigo (BPPV). Treatment of this disease are the relocation manoeuvres. Although these manoeuvres are effective in primary care (PC), they are not done routinely. Attention to other causes of vertigo in PC also has a wide margin for improvement. Objectives: To verify the effectiveness of a blended course in PC to improve adherence to clinical practice guidelines. Design: randomized community trial, by clusters (CG / IG), multicenter and open, taking as unit of allocation the primary care team (PCT). The professionals of the PCT that are in IG would receive the training at the beginning of the study and those of the control group will be offered after the conclusion of the same. Scope: 20 PCT (10 per group) selected from the "Costa de Ponent" Primary Care Directorate of the Catalan Health Institute. Variables: The outcome variables will be: Diagnostic records (proportion of nonspecific diagnoses such as dizziness and vertigo, with respect to specific diagnoses such as BPPV, vestibular neuritis); Derivations to otorhinolaryngologist (ENT) and neurologist; Prescription of antivertiginous medications and Number of days off work caused by vertigo-related illnesses during the study period. Other study variables will be characteristics of the professionals (age, sex) and centers (teachers, number of tutors, rural / urban). All the variables will be collected in an aggregated form by computerized data download during the year following the training intervention in the PCT. Statistical analysis: Following the CONSORT Cluster Guide, the baseline comparability of the two study groups will be analyzed to analyze the homogeneity. Descriptive statistics of all the baseline variables will be carried out and, the differences between groups in the post-intervention outcome variables will be evaluated through the t-test. In the IG, a multivariate logistic regression model will identify response patterns based on the baseline variables of professionals and centers. Conclusions: Positive results of the study could imply a paradigm shift in the approach to vertigo in primary care, which would be easy to extend to other areas since the most important part of the training course will be done online.

ELIGIBILITY:
Inclusion Criteria:

* 20 randomized primary care teams out of the 56 that make up the "Costa de Ponent" Primary Care Department that serve a population of 1.3 million people.

Exclusion Criteria:

* Primary care teams in which> 60% of their professionals have received a course on vertigo in the last 5 years will be excluded.
* Primary care teams who are not interested in participating in the study will be excluded

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic records | one year
  proportion of nonspecific diagnoses such as dizziness and vertigo, with respect to specific diagnoses such as BPPV, vestibular neuritis

SECONDARY OUTCOMES:
Derivations to otorhinolaryngologist (ENT) and neurologist | one year
  Number of referrals made during the study period
Prescription of antivertiginous medications | One year
  Number of prescriptions of betahistine, sulpiride, dimenhydrinate made during the study period
Days off work | One year
  Number of days off work caused by vertigo-related illnesses during the study period

CONTACTS AND LOCATIONS:
Overall Officials: José L Ballve, MD, PHD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina

REFERENCES:
- [Derived] Patino JEP, Moreno JLB, Matos YR, Ortega JA, Puertolas OC, Munoz RC, Balboa IV, Compta XG, Agudelo OLA, Munoz SC, Rodriguez VM, Cortes AN, Rodriguez EP. Effectiveness of a training intervention to improve the management of vertigo in primary care: a multicentre cluster-randomised trial, VERTAP. Trials. 2022 Jul 29;23(1):608. doi: 10.1186/s13063-022-06548-7. PMID 35906606